CLINICAL TRIAL: NCT02622321
Title: A Randomized, Multicenter, Open-Label, Phase III Clinical Trial to Evaluate the Efficacy, Safety, and Pharmacokinetics of Prophylactic Emicizumab Versus no Prophylaxis in Hemophilia A Patients With Inhibitors
Brief Title: A Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of Prophylactic Emicizumab Versus no Prophylaxis in Hemophilia A Participants With Inhibitors
Acronym: HAVEN 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Chugai Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BH29884; 2015-002866-21 (EudraCT Number)
Expanded Access: NCT03154437 (Approved for marketing)
Record Dates: First submitted 2015-12-02; First posted 2015-12-04 (Estimated); Results first posted 2017-11-24 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-05

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — emicizumab; recombinant FVIIa; anti-inhibitor coagulant complex

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm A: 1.5 mg/kg Emicizumab QW (Experimental): Participants who were receiving episodic treatment with bypassing agents prior to study entry and were randomized to study Arm A started to receive emicizumab prophylaxis. Emicizumab was administered at a loading dose of 3 milligrams per kilogram (mg/kg) once a week (QW) subcutaneously (SC) for the first 4 weeks followed by a maintenance dose of 1.5 mg/kg emicizumab QW SC up to the end of study. Participants continued to receive bypassing agent therapy to treat any breakthrough bleeds.
  Interventions: Drug: Emicizumab; Drug: rFVIIa; Drug: aPCC
- Arm B (Control): No Prophylaxis, Then Emicizumab (Active Comparator): Participants who were receiving episodic treatment with bypassing agents prior to study entry and were randomized to study Arm B continued with their prior episodic treatment regimen for the first 24 weeks of the study; they did not receive emicizumab prophylaxis during that time. After completing at least 24 weeks on study, participants in Arm B were allowed to switch to emicizumab prophylaxis (as described for Arm A) up to the end of study. Participants continued to receive bypassing agent therapy to treat any breakthrough bleeds.
  Interventions: Drug: Emicizumab; Drug: rFVIIa; Drug: aPCC
- Arm C: 1.5 mg/kg Emicizumab QW (Experimental): Participants who were receiving prophylactic bypassing agents prior to study entry were enrolled in Arm C to receive prophylactic emicizumab. Emicizumab was administered at a loading dose of 3 mg/kg QW SC for the first 4 weeks followed by a maintenance dose of 1.5 mg/kg emicizumab QW SC up to the end of study. Participants continued to receive bypassing agent therapy to treat any breakthrough bleeds.
  Interventions: Drug: Emicizumab; Drug: rFVIIa; Drug: aPCC
- Arm D: 1.5 mg/kg Emicizumab QW (Experimental): Participants who were either: 1) Receiving episodic bypassing agents prior to study entry but were unable to enroll in Arms A or B; or 2) Receiving bypassing agent prophylaxis prior to study entry but were unable to enroll in Arm C, were enrolled in Arm D to receive emicizumab prophylaxis. Emicizumab was administered at a loading dose of 3 mg/kg QW SC for the first 4 weeks followed by a maintenance dose of 1.5 mg/kg emicizumab QW SC up to the end of study. Participants continued to receive bypassing agent therapy to treat any breakthrough bleeds.
  Interventions: Drug: Emicizumab; Drug: rFVIIa; Drug: aPCC

INTERVENTIONS:
Drug: Emicizumab — Emicizumab will be administered at a loading dose of 3 milligrams per kilogram per week (mg/kg/week) subcutaneously (SC) for the first 4 weeks followed by a maintenance dose of 1.5 mg/kg/week SC up to the end of study. After at least 24 weeks on prophylactic emicizumab, individuals who experience suboptimal bleeding control on emicizumab (according to protocol-defined criteria) will have the opportunity to increase their dose to 3 mg/kg weekly.
  Other Names: Hemlibra; RO5534262; RG6013; ACE910
Drug: rFVIIa — Participants will continue to receive rFVIIa.
  Other Names: NovoSeven®
Drug: aPCC — Participants will continue to receive aPCC.
  Other Names: Factor Eight Inhibitor Bypassing Activity (FEIBA®)

SUMMARY:
This multicenter, open-label study will evaluate the safety, efficacy and pharmacokinetics of prophylactic emicizumab treatment in participants previously treated with episodic or prophylactic bypassing agents. Episodic bypassing agent participants will be randomized in a 2:1 fashion to receive emicizumab prophylaxis (Arm A) versus no prophylaxis (Arm B) and will be stratified across Arms A and B according to the number of bleeds they experienced over the last 24 weeks prior to study entry (less than [<] 9 or greater than or equal to [>/=] 9 bleeds); Arm B participants will have the opportunity to switch to emicizumab prophylaxis after at least 24 weeks on-study. Prophylactic bypassing agent participants will switch to emicizumab prophylaxis (Arm C) from the start of the trial; enrollment will be extended for 24 weeks after the last participant has enrolled in Arms A or B or until approximately 50 participants have enrolled in Arm C, whichever occurs first. Episodic bypassing agent participants who previously participated in the non-interventional study BH29768 (NCT02476942) who were unable to enroll in Arms A or B, or participants on prophylactic bypassing agents who were unable to enroll in Arm C, prior to their closure will have the opportunity to enroll in Arm D. Like participants in Arms A and C, Arm D participants will receive emicizumab prophylaxis from the start of the trial. All participants will continue to receive episodic bypassing agent therapy to treat breakthrough bleeds, preferably with recombinant activated factor VII (rFVIIa).

ELIGIBILITY:
Inclusion Criteria:

* Body weight >/= 40 kilograms (kg) at the time of screening
* Diagnosis of congenital hemophilia A of any severity and documented history of high-titer inhibitor ( that is [i.e.], >/= 5 Bethesda Units [BU])
* Documentation of treatment with episodic or prophylactic bypassing agents for at least the last 24 weeks
* >/= 6 bleeds in the last 24 weeks prior to screening (if on an episodic bypassing agent regimen) or >/=2 bleeds in the last 24 weeks prior to screening (if on a prophylactic bypassing agent regimen)
* Adequate hematologic, hepatic and renal function
* For women who are not postmenopausal or surgically sterile: agreement to remain abstinent or use single or combined highly effective contraceptive methods

Exclusion Criteria:

* Participants with inherited or acquired bleeding disorder other than hemophilia A
* Participants with ongoing (or plan to receive during the study) immune tolerance induction therapy or prophylaxis with Factor VIII (FVIII), with the exception of participants who have received a treatment regimen of FVIII prophylaxis with concurrent bypassing agent prophylaxis
* Previous (in the past 12 months) or current treatment for thromboembolic disease (with the exception of previous catheter-associated thrombosis for which antithrombotic treatment is not currently ongoing) or current signs of thromboembolic disease
* Participants with other conditions (for example [e.g.], certain autoimmune diseases) that may increase the risk of bleeding or thrombosis
* History of clinically significant hypersensitivity associated with monoclonal antibody therapies or components of the emicizumab injection
* Known human immunodeficiency virus (HIV) infection with cluster of differentiation 4 (CD4) count < 200 cells per microliter (cells/mcL) within 24 weeks prior to screening
* Use of systemic immunomodulators (e.g., interferon or rituximab) at enrolment or planned use during the study, with the exception of antiretroviral therapy
* Participants who are at high risk for thrombotic microangiopathy (TMA; e.g., have a previous medical or family history of TMA), in the investigator's judgment
* Concurrent disease, treatment, or abnormality in clinical laboratory tests that could interfere with the conduct of the study or that would, in the opinion of the investigator or Sponsor, preclude the participant's safe participation in and completion of the study or interpretation of the study results
* Planned surgery (excluding minor procedures such as tooth extraction or incision and drainage) during the study
* Receipt of emicizumab in a prior investigational study; An investigational drug to treat or reduce the risk of hemophilic bleeds within 5 half-lives of last drug administration; A non-hemophilia-related investigational drug within last 30 days or 5 half-lives, whichever is shorter; An investigational drug concurrently
* Unwillingness to use highly effective contraception methods for the specified duration in the protocol (females only, unless required otherwise by the local health authority)
* Clinically significant abnormality on screening evaluations or laboratory tests that, in the opinion of the investigator, may pose an additional risk in administering study drug to the participant
* Pregnancy or lactation, or intent to become pregnant during the study

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2015-11-18 (Actual); Primary Completion 2016-10-25 (Actual); Study Completion 2020-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (44):
- United States (11):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Santa Monica Oncology Center, Santa Monica, California
  - University of Colorado Denver, Children's Hospital, Aurora, Colorado
  - Winship Cancer Institute, Atlanta, Georgia
  - Boston Childrens Hospital, Boston, Massachusetts
  - Children's Hospital of Michigan; Pediatrics, Detroit, Michigan
  - Cornell Univ Medical College; Hematology-Oncolog, New York, New York
  - Oregon Health & Science Uni ; Dept of Pediatrics, Portland, Oregon
  - Pennsylvania State Hershey Medical Center; Division of Hematology/Oncology, H046, Hershey, Pennsylvania
  - Univ of TX Health Science Ctr; Gulf States Hemo and Throm Ctr, Houston, Texas
  - Bloodworks Northwest (formerly Puget Sound Blood Center); Hemophilia, Seattle, Washington
- Australia (2):
  - Royal Prince Alfred Hospital; Haematology, Camperdown, New South Wales
  - The Alfred Hospital, Melbourne; Thrombosis and Haemostasis Unit, Melbourne, Victoria
- ICIC, San José, Costa Rica
- France (4):
  - Hopital Cardio-vasculaire Louis Pradel; Hemostase clinique, Bron
  - CH de Bicetre; Centre de Traitement d' Hemophilie, Le Kremlin-Bicêtre
  - Hopital Cardiologique; Hematologie B, Lille
  - Groupe Hospitalier Necker Enfants Malades, Paris
- Germany (3):
  - Universitätsklinikum Bonn; Institut für Experimentelle Hämatologie und Transfusionsmedizin, Bonn
  - CTC North GmbH & Co. KG am Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Hämophilie-Zentrum Rhein Main GmbH, Mörfelden-Walldorf
- Italy (2):
  - IRCCS Ca' Granda Ospedale Maggiore Policlinico; Centro Emofilia e Trombosi "Angelo Bianchi e Bonomi", Milan, Lombardy
  - AOU Careggi; SOD Malattie Emorragiche, Florence, Tuscany
- Japan (7):
  - Nagoya University Hospital, Aichi
  - Hiroshima University Hospital, Hiroshima
  - Hyogo College of Medicine Hospital, Hyōgo
  - St. Marianna University School of Medicine Hospital, Kanagawa
  - Hospital of the University of Occupational and Environmental Health,Japan, Kitakyushu-shi
  - Nara Medical University Hospital, Nara
  - Tokyo Medical University Hospital, Tokyo
- Auckland City Hospital; Auckland Haemophilia Centre, Auckland, New Zealand
- Poland (4):
  - Uniwersyteckie Centrum Kliniczne; Klinika Hematologii i Transplantologii, Gdansk
  - SPSK Nr1 Klinika Hematoo&Transpl.Szpiku, Lublin
  - ALVAMED Lekarskie Gabinety Specjalistyczne, Poznan
  - Instytut Hematologii i Transfuzjologii; Klinika Zaburzeń Hemostazy i Chorób Wewnętrznych, Warsaw
- Charlotte Maxeke Johannesburg Hospital; Haemophilia Comprehensive Care Center, Johannesburg, South Africa
- Severance Hospital, Seoul, South Korea
- Spain (3):
  - Hospital Universitario la Paz; Servicio de Hematologia, Madrid
  - Hospital Universitario Virgen del Rocio; Servicio de Hematologia, Seville
  - Hospital Universitario la Fe; Servicio de Hematologia, Valencia
- National Taiwan Uni Hospital, Taipei, Taiwan
- United Kingdom (3):
  - Cardiff and Vale NHS Trust, Cardiff
  - St Thomas' Hospital; Haemostasis & Thromboisis Centre, London
  - Oxford University Hospitals NHS Trust - Churchill Hospital, Oxford

REFERENCES:
- [Derived] Kruse-Jarres R, Peyvandi F, Oldenburg J, Chang T, Chebon S, Doral MY, Croteau SE, Lambert T, Kempton CL, Pipe SW, Ko RH, Trzaskoma B, Dhalluin C, Bienz NS, Niggli M, Lehle M, Paz-Priel I, Young G, Jimenez-Yuste V. Surgical outcomes in people with hemophilia A taking emicizumab prophylaxis: experience from the HAVEN 1-4 studies. Blood Adv. 2022 Dec 27;6(24):6140-6150. doi: 10.1182/bloodadvances.2022007458. PMID 35939785
- [Derived] Oldenburg J, Mahlangu JN, Kim B, Schmitt C, Callaghan MU, Young G, Santagostino E, Kruse-Jarres R, Negrier C, Kessler C, Valente N, Asikanius E, Levy GG, Windyga J, Shima M. Emicizumab Prophylaxis in Hemophilia A with Inhibitors. N Engl J Med. 2017 Aug 31;377(9):809-818. doi: 10.1056/NEJMoa1703068. Epub 2017 Jul 10. PMID 28691557

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 113 participants were enrolled in this study: 109 participants prior to the primary completion date plus a further 4 participants to Arm D of the study after the primary completion date. Participants in Arm A and Arm B were randomized in a 2:1 ratio; participants in Arm C and Arm D were enrolled without randomization.
Period: Overall Study
Arm/Group | Arm A: 1.5 mg/kg Emicizumab QW | Arm B (Control): No Prophylaxis, Then Emicizumab | Arm C: 1.5 mg/kg Emicizumab QW | Arm D: 1.5 mg/kg Emicizumab QW
Started | 35 | 18 | 49 | 11
Received at Least One Dose of Treatment (Safety Population) | 34 (1 participant withdrew prior to study Day 1.) | 18 | 49 | 11
Completed 24 Weeks in the Study | 31 | 18 (After 24 weeks, all 18 participants in Arm B switched to receive emicizumab prophylaxis.) | 49 | 11
Dose Up-Titrated to 3 mg/kg QW | 2 | 0 | 3 | 2
Completed | 32 | 18 | 48 | 11
Not Completed | 3 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 1 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: 1.5 mg/kg Emicizumab QW | Arm B (Control): No Prophylaxis, Then Emicizumab | Arm C: 1.5 mg/kg Emicizumab QW | Arm D: 1.5 mg/kg Emicizumab QW | Total
Number analyzed (Participants) | 35 | 18 | 49 | 11 | 113
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.8 (13.9) | 37.2 (13.7) | 25.6 (16.8) | 39.0 (16.1) | 31.9 (16.2)
Age, Customized [Count of Participants; unit: Participants]
  Adolescents (12-17 years) | 4 | 2 | 26 | 0 | 32
  Adults (18-64 years) | 30 | 15 | 21 | 10 | 76
  Elderly (65-84 years) | 1 | 1 | 2 | 1 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 35 | 18 | 49 | 11 | 113
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 12 | 1 | 18
  Not Hispanic or Latino | 31 | 17 | 37 | 10 | 95
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 10 | 3 | 8 | 0 | 21
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 1
  Black or African American | 4 | 4 | 3 | 0 | 11
  White | 21 | 10 | 33 | 11 | 75
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 4 | 0 | 4
Number of Participants by the Number of Bleeds (<9 or ≥9) in the Last 24 Weeks Prior to Study Entry [Count of Participants; unit: Participants]
  <9 Bleeds | 11 | 5 | 23 | 6 | 45
  ≥9 Bleeds | 24 | 13 | 26 | 5 | 68

OUTCOME MEASURES:

1. Primary Outcome: Model-Based Annualized Bleed Rate (ABR) for Treated Bleeds, Arm A: Emicizumab Versus Arm B: No Prophylaxis
Description: The number of treated bleeds over the efficacy period was assessed as an annualized bleed rate (ABR) using a negative binomial (NB) regression model, which accounts for different follow-up times. Treated bleeds were defined as a bleed that was directly followed by a hemophilia medication reported to be a "treatment for bleed". The 72-hour rule was implemented: two bleeds of the same type and at the same anatomical location were counted as one bleed if the second bleed occurred within 72 hours from the last treatment for the first bleed. Bleeds due to surgery/procedure were excluded. For participants whose dose was up-titrated, the efficacy period ended the day before the first day on the up-titrated dose.
Time Frame: From Baseline up to 24 weeks (median [min-max] efficacy observation periods in Arm A vs. Arm B: 29.29 [0.1-48.9] weeks vs. 24.14 [23.0-26.0] weeks)
Population: Intent-to-treat (ITT) population defined as all participants who were randomized to Arm A or Arm B.
Measure: Number (95% Confidence Interval); unit: treated bleeds per year
Groups:
- Arm B (Control): No Prophylaxis: Participants who were receiving episodic treatment with bypassing agents prior to study entry and were randomized to study Arm B continued with their prior episodic treatment regimen for the first 24 weeks of the study; they did not receive emicizumab prophylaxis during that time. After completing at least 24 weeks on study, participants in Arm B were allowed to switch to emicizumab prophylaxis (as described for Arm A) up to the end of study. Participants continued to receive bypassing agent therapy to treat any breakthrough bleeds.
Arm/Group | Arm A: 1.5 mg/kg Emicizumab QW | Arm B (Control): No Prophylaxis
Number analyzed (Participants) | 35 | 18
treated bleeds per year | 2.9 [1.69 to 5.02] | 23.3 [12.33 to 43.89]
Statistical Analysis 1: Comparison: Arm A: 1.5 mg/kg Emicizumab QW vs Arm B (Control): No Prophylaxis; Analysis was performed using an NB regression model, which accounted for different follow-up times, with the participant's number of bleeds as a function of randomization and the time that each participant stays in the study included as an offset in the model. The model also included the number of bleeds (less than [<] 9 or greater than or equal to [>/=] 9) in the last 24 weeks prior to study entry as a stratification factor in the randomization; Test type: Superiority or Other; p < 0.0001, Stratified Wald Test — Statistical significance was controlled at a two-sided alpha level of 0.05 based on a Wald testing procedure; ABR Ratio = 0.13, 95% CI 2-sided [0.057 to 0.277]

2. Secondary Outcome: Model-Based Annualized Bleed Rate (ABR) for All Bleeds, Arm A: Emicizumab Versus Arm B: No Prophylaxis
Description: The number of all bleeds over the efficacy period was assessed as an annualized bleed rate (ABR) using a negative binomial (NB) regression model, which accounts for different follow-up times. All bleeds included both treated bleeds (with coagulation factors) and non-treated bleeds. The 72-hour rule was implemented: two bleeds of the same type and at the same anatomical location were counted as one bleed if the second bleed occurred within 72 hours from the last treatment for the first bleed. Bleeds due to surgery/procedure were excluded. For participants whose dose was up-titrated, the efficacy period ended the day before the first day on the up-titrated dose.
Time Frame: as for outcome 1
Population: ITT population: all participants who were randomized to Arm A or Arm B.
Measure: Number (95% Confidence Interval); unit: all bleeds per year
Arm/Group | Arm A: 1.5 mg/kg Emicizumab QW | Arm B (Control): No Prophylaxis
Number analyzed (Participants) | 35 | 18
all bleeds per year | 5.5 [3.58 to 8.60] | 28.3 [16.79 to 47.76]
Statistical Analysis 1: Comparison: Arm A: 1.5 mg/kg Emicizumab QW vs Arm B (Control): No Prophylaxis; Analysis was performed using an NB regression model, which accounted for different follow-up times, with the participant's number of bleeds as a function of randomization and the time that each participant stays in the study included as an offset in the model. The model also included the number of bleeds (<9 or >/=9) in the last 24 weeks prior to study entry as a stratification factor in the randomization; Test type: Superiority or Other; p < 0.0001, Stratified Wald Test — Statistical significance was controlled at a two-sided alpha level of 0.05 based on a Wald testing procedure; ABR Ratio = 0.20, 95% CI 2-sided [0.102 to 0.375]

3. Secondary Outcome: Intra-Participant Comparison of the Model-Based Annualized Bleed Rate (ABR) for All Bleeds in Arm A: Emicizumab Versus Previous Episodic Bypassing Agents
Description: This was an intra-participant comparison of the annualized bleed rates (ABRs) for all bleeds in Arm A participants who had previously received episodic bypassing agents during the non-interventional study (NIS) BH29768 (NCT02476942) (Arm A NIS) prior to entry in this study versus emicizumab prophylaxis during this study (Arm A). The number of all bleeds over the efficacy period was assessed as an ABR using a negative binomial (NB) regression model, which accounts for different follow-up times. All bleeds included both treated bleeds (with coagulation factors) and non-treated bleeds. The 72-hour rule was implemented: two bleeds of the same type and at the same anatomical location were counted as one bleed if the second bleed occurred within 72 hours from the last treatment for the first bleed. Bleeds due to surgery/procedure were excluded. For participants whose dose was up-titrated, the efficacy period ended the day before the first day on the up-titrated dose.
Time Frame: Median [min-max] efficacy observation periods: for Arm A, 1.5 mg/kg Emicizumab QW: 30.86 [0.1-48.9] weeks; for Arm A (NIS), Previous Episodic Bypassing Agents: 21.14 [10.6-33.9] weeks
Population: Arm A NIS population included all Arm A participants who participated in NIS BH29768 before study entry and received episodic bypassing agents during NIS BH29768.
Measure: Number (95% Confidence Interval); unit: all bleeds per year
Groups:
- Arm A (NIS): Previous Episodic Bypassing Agents: This arm includes data collected before entry into this study (assessed prospectively in a non-interventional study [NIS]) from Arm A participants who previously participated in NIS BH29768 (NCT02476942) and had received episodic bypassing agents during the NIS.
Arm/Group | Arm A: 1.5 mg/kg Emicizumab QW | Arm A (NIS): Previous Episodic Bypassing Agents
Number analyzed (Participants) | 24 | 24
all bleeds per year | 4.1 [2.10 to 8.02] | 37.7 [28.40 to 50.04]
Statistical Analysis 1: Comparison: Arm A: 1.5 mg/kg Emicizumab QW vs Arm A (NIS): Previous Episodic Bypassing Agents; This intra-participant comparison of ABR for all bleeds was performed using an NB regression model; Test type: Superiority or Other; p < 0.0001, Non-Stratified Wald Test — Statistical significance was controlled at a two-sided alpha level of 0.05 based on a Wald testing procedure; ABR Ratio = 0.11, 95% CI 2-sided [0.055 to 0.218]

4. Secondary Outcome: Intra-Participant Comparison of the Model-Based Annualized Bleed Rate (ABR) for Treated Bleeds in Arm A: Emicizumab Versus Previous Episodic Bypassing Agents
Description: This was an intra-participant comparison of the ABRs for treated bleeds in Arm A participants who had previously received episodic bypassing agents during the non-interventional study (NIS) BH29768 (NCT02476942) (Arm A NIS) prior to entry in this study versus emicizumab prophylaxis during this study (Arm A). The number of treated bleeds over the efficacy period was assessed as an ABR using a negative binomial (NB) regression model, which accounts for different follow-up times. Treated bleeds were defined as a bleed that was directly followed by a hemophilia medication reported to be a "treatment for bleed". The 72-hour rule was implemented: two bleeds of the same type and at the same anatomical location were counted as one bleed if the second bleed occurred within 72 hours from the last treatment for the first bleed. Bleeds due to surgery/procedure were excluded. For participants whose dose was up-titrated, efficacy period ended the day before the first day on the up-titrated dose.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: treated bleeds per year
Arm/Group | Arm A: 1.5 mg/kg Emicizumab QW | Arm A (NIS): Previous Episodic Bypassing Agents
Number analyzed (Participants) | 24 | 24
treated bleeds per year | 1.7 [0.71 to 4.06] | 21.6 [15.40 to 30.22]
Statistical Analysis 1: Comparison: Arm A: 1.5 mg/kg Emicizumab QW vs Arm A (NIS): Previous Episodic Bypassing Agents; This intra-participant comparison of ABR for treated bleeds was performed using an NB regression model; Test type: Superiority or Other; p < 0.0001, Non-Stratified Wald Test — Statistical significance was controlled at a two-sided alpha level of 0.05 based on a Wald testing procedure; ABR Ratio = 0.08, 95% CI 2-sided [0.031 to 0.198]

5. Secondary Outcome: Model-Based Annualized Bleed Rate (ABR) for Treated Joint Bleeds, Arm A: Emicizumab Versus Arm B: No Prophylaxis
Description: The number of treated joint bleeds over the efficacy period was assessed as an ABR using a negative binomial (NB) regression model, which accounts for different follow-up times. Treated joint bleeds were defined as treated bleeds in a joint associated with unusual sensation (aura) in a joint, in combination with another symptom: swelling/warmth, pain/decreased range of motion (RoM), or difficulty moving the joint. Bleeds due to surgery/procedure were excluded.
Time Frame: as for outcome 1
Population: ITT population: all participants who were randomized to Arm A or Arm B.
Measure: Number (95% Confidence Interval); unit: treated joint bleeds per year
Arm/Group | Arm A: 1.5 mg/kg Emicizumab QW | Arm B (Control): No Prophylaxis
Number analyzed (Participants) | 35 | 18
treated joint bleeds per year | 0.8 [0.26 to 2.20] | 6.7 [1.99 to 22.42]
Statistical Analysis 1: Comparison: Arm A: 1.5 mg/kg Emicizumab QW vs Arm B (Control): No Prophylaxis; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0050, Stratified Wald Test — Statistical significance was controlled at a two-sided alpha level of 0.05 based on a Wald testing procedure; ABR Ratio = 0.11, 95% CI 2-sided [0.025 to 0.520]

6. Secondary Outcome: Intra-Participant Comparison of the Model-Based Annualized Bleed Rate (ABR) for All Bleeds in Arm C: Emicizumab Versus Previous Prophylactic Bypassing Agents
Description: This was an intra-participant comparison of the annualized bleed rates (ABRs) for all bleeds in Arm C participants who had previously received prophylactic bypassing agents during the non-interventional study (NIS) BH29768 (NCT02476942) (Arm C NIS) prior to entry in this study versus emicizumab prophylaxis during this study (Arm C). The number of all bleeds over the efficacy period was assessed as an ABR using a negative binomial (NB) regression model, which accounts for different follow-up times. All bleeds included both treated bleeds (with coagulation factors) and non-treated bleeds. The 72-hour rule was implemented: two bleeds of the same type and at the same anatomical location were counted as one bleed if the second bleed occurred within 72 hours from the last treatment for the first bleed. Bleeds due to surgery/procedure were excluded. For participants whose dose was up-titrated, the efficacy period ended the day before the first day on the up-titrated dose.
Time Frame: Median [min-max] efficacy observation periods: for Arm C, 1.5 mg/kg Emicizumab QW: 30.14 [6.9-45.3] weeks; for Arm C (NIS), Previous Prophylactic Bypassing Agents: 32.14 [8.1-49.3] weeks
Population: Arm C NIS population included all Arm C participants who participated in NIS BH29768 before study entry and received prophylactic bypassing agents during NIS BH29768.
Measure: Number (95% Confidence Interval); unit: all bleeds per year
Groups:
- Arm C (NIS): Previous Prophylactic Bypassing Agents: This arm includes data collected before entry into this study (assessed prospectively in a non-interventional study [NIS]) from Arm C participants who previously participated in NIS BH29768 (NCT02476942) and had received prophylactic bypassing agents during the NIS.
Arm/Group | Arm C: 1.5 mg/kg Emicizumab QW | Arm C (NIS): Previous Prophylactic Bypassing Agents
Number analyzed (Participants) | 24 | 24
all bleeds per year | 5.5 [2.98 to 10.26] | 24.3 [18.11 to 32.67]
Statistical Analysis 1: Comparison: Arm C: 1.5 mg/kg Emicizumab QW vs Arm C (NIS): Previous Prophylactic Bypassing Agents; This intra-participant comparison of ABR for all bleeds was performed using an NB regression model; Test type: Superiority or Other; p < 0.0001, Non-Stratified Wald Test — Statistical significance was controlled at a two-sided alpha level of 0.05 based on a Wald testing procedure; ABR Ratio = 0.23, 95% CI 2-sided [0.119 to 0.435]

7. Secondary Outcome: Intra-Participant Comparison of the Model-Based Annualized Bleed Rate (ABR) for Treated Bleeds in Arm C: Emicizumab Versus Previous Prophylactic Bypassing Agents
Description: This was an intra-participant comparison of the ABRs for treated bleeds in Arm C participants who had previously received bypassing agent prophylaxis during the non-interventional study (NIS) BH29768 (NCT02476942) (Arm C NIS) prior to entry in this study versus emicizumab prophylaxis during this study (Arm C). The number of treated bleeds over the efficacy period was assessed as an ABR using a negative binomial (NB) regression model, which accounts for different follow-up times. Treated bleeds were defined as a bleed that was directly followed by a hemophilia medication reported to be a "treatment for bleed". The 72-hour rule was implemented: two bleeds of the same type and at the same anatomical location were counted as one bleed if the second bleed occurred within 72 hours from the last treatment for the first bleed. Bleeds due to surgery/procedure were excluded. For participants whose dose was up-titrated, efficacy period ended the day before the first day on the up-titrated dose.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: treated bleeds per year
Groups:
- Arm Cnis: Previous Prophylactic Bypassing Agents: This arm includes data collected before entry into this study (assessed prospectively in a non-interventional study [NIS]) from Arm C participants who previously participated in NIS BH29768 (NCT02476942) and had received prophylactic bypassing agents (rFVIIa or/and aPCC) during the NIS BH29768.
Arm/Group | Arm C: 1.5 mg/kg Emicizumab QW | Arm Cnis: Previous Prophylactic Bypassing Agents
Number analyzed (Participants) | 24 | 24
treated bleeds per year | 3.3 [1.33 to 8.08] | 15.7 [11.08 to 22.29]
Statistical Analysis 1: Comparison: Arm C: 1.5 mg/kg Emicizumab QW vs Arm Cnis: Previous Prophylactic Bypassing Agents; This intra-participant comparison of ABR for treated bleeds was performed using an NB regression model; Test type: Superiority or Other; p = 0.0003, Non-Stratified Wald Test — Statistical significance was controlled at a two-sided alpha level of 0.05 based on a Wald testing procedure; ABR Ratio = 0.21, 95% CI 2-sided [0.089 to 0.486]

8. Secondary Outcome: Model-Based Annualized Bleed Rate (ABR) for Treated Spontaneous Bleeds, Arm A: Emicizumab Versus Arm B: No Prophylaxis
Description: The number of treated spontaneous bleeds over the efficacy period was assessed as an annualized bleed rate (ABR) using a negative binomial (NB) regression model, which accounts for different follow-up times. Treated spontaneous bleeds were defined as treated (with coagulation factors) bleeds with no known contributing factor (e.g., trauma, surgery). The 72-hour rule was implemented: two bleeds of the same type and at the same anatomical location were counted as one bleed if the second bleed occurred within 72 hours from the last treatment for the first bleed. Bleeds due to surgery/procedure were excluded. For participants whose dose was up-titrated, the efficacy period ended the day before the first day on the up-titrated dose.
Time Frame: as for outcome 1
Population: ITT population: all participants who were randomized to Arm A or Arm B.
Measure: Number (95% Confidence Interval); unit: treated spontaneous bleeds per year
Arm/Group | Arm A: 1.5 mg/kg Emicizumab QW | Arm B (Control): No Prophylaxis
Number analyzed (Participants) | 35 | 18
treated spontaneous bleeds per year | 1.3 [0.73 to 2.19] | 16.8 [9.94 to 28.30]
Statistical Analysis 1: Comparison: Arm A: 1.5 mg/kg Emicizumab QW vs Arm B (Control): No Prophylaxis; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, Stratified Wald Test — Statistical significance was controlled at a two-sided alpha level of 0.05 based on a Wald testing procedure; ABR Ratio = 0.08, 95% CI 2-sided [0.037 to 0.154]

9. Secondary Outcome: Model-Based Annualized Bleed Rate (ABR) for Treated Target Joint Bleeds, Arm A: Emicizumab Versus Arm B: No Prophylaxis
Description: The number of treated target joint bleeds over the efficacy period was assessed as an annualized bleed rate (ABR) using a negative binomial (NB) regression model, which accounts for different follow-up times. Treated target joint bleeds included treated (with coagulation factors) joint bleeds in a target joint, defined as a joint in which greater than or equal to (>/=) 3 treated joint bleeds occurred during the last 24 weeks prior to study entry. The 72-hour rule was implemented: two bleeds of the same type and at the same anatomical location were counted as one bleed if the second bleed occurred within 72 hours from the last treatment for the first bleed. Bleeds due to surgery/procedure were excluded. For participants whose dose was up-titrated, the efficacy period ended the day before the first day on the up-titrated dose.
Time Frame: as for outcome 1
Population: ITT population: all participants who were randomized to Arm A or Arm B.
Measure: Number (95% Confidence Interval); unit: treated target joint bleeds per year
Arm/Group | Arm A: 1.5 mg/kg Emicizumab QW | Arm B (Control): No Prophylaxis
Number analyzed (Participants) | 35 | 18
treated target joint bleeds per year | 0.1 [0.03 to 0.58] | 3.0 [0.96 to 9.13]
Statistical Analysis 1: Comparison: Arm A: 1.5 mg/kg Emicizumab QW vs Arm B (Control): No Prophylaxis; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0002, Stratified Wald Test — Statistical significance was controlled at a two-sided alpha level of 0.05 based on a Wald testing procedure; ABR Ratio = 0.05, 95% CI 2-sided [0.009 to 0.227]

10. Secondary Outcome: Mean Calculated Annualized Bleed Rates (ABR) for Treated Bleeds, All Bleeds, Treated Spontaneous Bleeds, Treated Joint Bleeds, and Treated Target Joint Bleeds, Arm A: Emicizumab Versus Arm B: No Prophylaxis
Description: The number of bleeds over the efficacy period was calculated as: ABR = (number of bleeds/number of days during the efficacy period) x 365.25. Treated bleeds: a bleed for which coagulation factors were administered. All bleeds included both treated and non-treated bleeds. Treated spontaneous bleeds: treated bleeds with no known contributing factor (e.g., trauma, surgery). Treated joint bleeds: treated bleeds in a joint associated with unusual sensation (aura) in a joint, in combination with another symptom: swelling/warmth, pain/decreased range of motion (RoM), or difficulty moving the joint. Treated target joint bleeds: treated joint bleeds in a target joint, defined as a joint in which greater than or equal to (>/=) 3 treated joint bleeds occurred during the last 24 weeks prior to study entry. For all types of bleeds: the 72-hour rule was implemented, and bleeds due to surgery/procedure and bleeds after up-titration were excluded.
Time Frame: as for outcome 1
Population: ITT population: all participants who were randomized to Arm A or Arm B.
Measure: Mean (95% Confidence Interval); unit: bleeds per year
Arm/Group | Arm A: 1.5 mg/kg Emicizumab QW | Arm B (Control): No Prophylaxis
Number analyzed (Participants) | 35 | 18
bleeds per year
  Treated Bleeds | 3.5 [0.83 to 9.46] | 26.2 [17.17 to 38.37]
  All Bleeds | 6.3 [2.37 to 13.45] | 30.8 [20.89 to 43.76]
  Treated Spontaneous Bleeds | 1.5 [0.11 to 6.42] | 18.1 [10.74 to 28.57]
  Treated Joint Bleeds | 1.0 [0.03 to 5.57] | 8.1 [3.55 to 15.95]
  Treated Target Joint Bleeds | 0.4 [0.00 to 4.48] | 6.2 [2.32 to 13.34]

11. Secondary Outcome: Median Calculated Annualized Bleed Rates (ABR) for Treated Bleeds, All Bleeds, Treated Spontaneous Bleeds, Treated Joint Bleeds, and Treated Target Joint Bleeds, Arm A: Emicizumab Versus Arm B: No Prophylaxis
Description: as for outcome 10
Time Frame: as for outcome 1
Population: ITT population: all participants who were randomized to Arm A or Arm B.
Measure: Median (Inter-Quartile Range); unit: bleeds per year
Arm/Group | Arm A: 1.5 mg/kg Emicizumab QW | Arm B (Control): No Prophylaxis
Number analyzed (Participants) | 35 | 18
bleeds per year
  Treated Bleeds | 0.0 [0.00 to 3.73] | 18.8 [12.97 to 35.08]
  All Bleeds | 2.0 [0.00 to 9.87] | 30.2 [18.26 to 39.37]
  Treated Spontaneous Bleeds | 0.0 [0.00 to 3.28] | 15.2 [6.64 to 30.44]
  Treated Joint Bleeds | 0.0 [0.00 to 0.00] | 1.0 [0.00 to 14.44]
  Treated Target Joint Bleeds | 0.0 [0.00 to 0.00] | 1.0 [0.00 to 6.52]

12. Secondary Outcome: Percentage of Participants With 0 Bleeds for Treated Bleeds, All Bleeds, Treated Spontaneous Bleeds, Treated Joint Bleeds, and Treated Target Joint Bleeds, Arm A: Emicizumab Versus Arm B: No Prophylaxis
Description: Treated bleeds: a bleed for which coagulation factors were administered. All bleeds included both treated and non-treated bleeds. Treated spontaneous bleeds: treated bleeds with no known contributing factor (e.g., trauma, surgery). Treated joint bleeds: treated bleeds in a joint associated with unusual sensation (aura) in a joint, in combination with another symptom: swelling/warmth, pain/decreased range of motion (RoM), or difficulty moving the joint. Treated target joint bleeds: treated joint bleeds in a target joint, defined as a joint in which greater than or equal to (>/=) 3 treated joint bleeds occurred during the last 24 weeks prior to study entry. For all types of bleeds: the 72-hour rule was implemented, and bleeds due to surgery/procedure and bleeds after up-titration were excluded.
Time Frame: as for outcome 1
Population: ITT population: all participants who were randomized to Arm A or Arm B.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: 1.5 mg/kg Emicizumab QW | Arm B (Control): No Prophylaxis
Number analyzed (Participants) | 35 | 18
Percentage of participants
  Treated Bleeds | 62.9 [44.9 to 78.5] | 5.6 [0.1 to 27.3]
  All Bleeds | 37.1 [21.5 to 55.1] | 5.6 [0.1 to 27.3]
  Treated Spontaneous Bleeds | 68.6 [50.7 to 83.1] | 11.1 [1.4 to 34.7]
  Treated Joint Bleeds | 85.7 [69.7 to 95.2] | 50.0 [26.0 to 74.0]
  Treated Target Joint Bleeds | 94.3 [80.8 to 99.3] | 50.0 [26.0 to 74.0]

13. Secondary Outcome: Hemophilia-Specific Quality of Life (Haem-A-QoL) Questionnaire Physical Health Score at Week 25 in Adult Participants (>/=18 Years Old), Arm A: Emicizumab Versus Arm B: No Prophylaxis
Description: Haem-A-QoL questionnaire has been developed and used in hemophilia A participants. As a hemophilia-specific questionnaire, this measure assesses very specific aspects of dealing with hemophilia. This questionnaire consists of items pertaining to 10 domains specific to living with hemophilia. The 10 domains are: physical health, sports and leisure, school and work, dealing with hemophilia, family planning, feeling, relationships, treatment, view of yourself, and outlook for the future. The total score for each domain range from 0 to 100 with lower scores reflective of better quality of life. Physical Health domain score is reported (range 0 to 100, with lower scores reflective of better physical health).
Time Frame: Week 25
Population: ITT population: all participants who were randomized to Arm A or Arm B. The number of participants analyzed is the number of adult participants (≥18 years old) in Arms A and B who responded to the questionnaire at Week 25.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A: 1.5 mg/kg Emicizumab QW | Arm B (Control): No Prophylaxis
Number analyzed (Participants) | 26 | 14
score on a scale | 30.19 (26.59) | 57.14 (23.35)
Statistical Analysis 1: Comparison: Arm A: 1.5 mg/kg Emicizumab QW vs Arm B (Control): No Prophylaxis; Actual number of participants included for inferential statistics in Arm A is 25. Means adjusted for covariates: baseline score, treatment group and treatment by baseline interaction arm. Analysis was performed using Analysis of Covariance (ANCOVA); Test type: Superiority or Other; p = 0.0029, ANCOVA — Statistical significance was controlled at a two-sided alpha level of 0.05; Adjusted Mean Difference = 21.55, 95% CI 2-sided [7.89 to 35.22]

14. Secondary Outcome: Haem-A-QoL Questionnaire Total Score at Week 25 in Adult Participants (>/=18 Years Old), Arm A: Emicizumab Versus Arm B: No Prophylaxis
Description: Haem-A-QoL questionnaire has been developed and used in hemophilia A participants. As a hemophilia-specific questionnaire, this measure assesses very specific aspects of dealing with hemophilia. This questionnaire consists of items pertaining to 10 domains specific to living with hemophilia. The 10 domains are: physical health, sports and leisure, school and work, dealing with hemophilia, family planning, feeling, relationships, treatment, view of yourself, and outlook for the future. The total score for each domain range from 0 to 100 with lower scores reflective of better quality of life. Haem-A-QoL Questionnaire Total Score is the average of the all domain scores and range from 0 to 100, with lower scores reflective of better quality of life.
Time Frame: Week 25
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A: 1.5 mg/kg Emicizumab QW | Arm B (Control): No Prophylaxis
Number analyzed (Participants) | 26 | 14
score on a scale | 26.465 (18.666) | 47.504 (17.435)
Statistical Analysis 1: Comparison: Arm A: 1.5 mg/kg Emicizumab QW vs Arm B (Control): No Prophylaxis; Actual number of participants included for inferential statistics in Arm A is 25. Means adjusted for covariates: baseline score, treatment group and treatment by baseline interaction arm; Test type: Superiority or Other; p = 0.0019, ANCOVA — Statistical significance was controlled at a two-sided alpha level of 0.05; Adjusted Mean Difference = 14.01, 95% CI 2-sided [5.56 to 22.45]

15. Secondary Outcome: European Quality of Life-5 Dimensions-5 Levels (EQ-5D-5L) Visual Analog Scale Score at Week 25, Arm A: Emicizumab Versus Arm B: No Prophylaxis
Description: EQ-5D-5L is a standardized, participant-rated questionnaire to assess health-related quality of life. The EQ-5D-5L includes 2 components: the EQ-5D-5L health state profile (descriptive system) and the EQ-5D-5L Visual Analog Scale. The Visual Analogue Scale is designed to rate the participant's current health state on a scale from 0 to 100, where 0 represents the worst imaginable health state and 100 represents the best imaginable health state.
Time Frame: Week 25
Population: ITT population: all participants who were randomized to Arm A or Arm B. The number of participants analyzed is the number of participants in Arms A and B who responded to the questionnaire at Week 25.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A: 1.5 mg/kg Emicizumab QW | Arm B (Control): No Prophylaxis
Number analyzed (Participants) | 30 | 16
score on a scale | 83.8 (12.9) | 76.4 (15.7)
Statistical Analysis 1: Comparison: Arm A: 1.5 mg/kg Emicizumab QW vs Arm B (Control): No Prophylaxis; Actual number of participants included for inferential statistics in Arm A is 29. Means adjusted for covariates: baseline score, treatment group and treatment by baseline interaction arm; Test type: Superiority or Other; p = 0.0171, ANCOVA — Statistical significance was controlled at a two-sided alpha level of 0.05; Adjusted Mean Difference = -9.72, 95% CI 2-sided [-17.62 to -1.82]

16. Secondary Outcome: EQ-5D-5L Index Utility Score at Week 25, Arm A: Emicizumab Versus Arm B: No Prophylaxis
Description: EQ-5D-5L is a standardized, participant-rated questionnaire to assess health-related quality of life. The EQ-5D-5L includes 2 components: the EQ-5D-5L health state profile (descriptive system) and the EQ-5D-5L Visual Analog Scale. The EQ-5D-5L health state profile is designed to record the participant's current health state in 5 domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Responses from the five domains are used to calculate a single utility index value ranging from 1 to 5, where 1 indicates better health state (no problems) and 5 indicates worst health state (confined to bed).
Time Frame: Week 25
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A: 1.5 mg/kg Emicizumab QW | Arm B (Control): No Prophylaxis
Number analyzed (Participants) | 30 | 16
score on a scale | 0.83 (0.22) | 0.60 (0.35)
Statistical Analysis 1: Comparison: Arm A: 1.5 mg/kg Emicizumab QW vs Arm B (Control): No Prophylaxis; [analysis description as in outcome 15, analysis 1]; Test type: Superiority or Other; p = 0.0014, ANCOVA — Statistical significance was controlled at a two-sided alpha level of 0.05; Adjusted Mean Difference = -0.16, 95% CI 2-sided [-0.25 to -0.07]

17. Secondary Outcome: Hemophilia-Specific Quality of Life - Short Form (Haemo-Qol-SF) Questionnaire Total Score at Baseline and Week 25 in Adolescent Participants (12-17 Years Old)
Description: The Haemo-QoL-SF contains 35 items, which cover nine domains considered relevant for the children's health-related quality of life (physical health, feelings, view of yourself, family, friends, other people, sports and school, dealing with hemophilia and treatment). Items are rated with five respective response options: never, seldom, sometimes, often, and always. Haemo-QoL-SF total score range from 0 to 100, where lower scores reflect better health-related quality of life. Baseline was defined as the last assessment prior to treatment. Because participants in Arm B switched from episodic bypassing agents to start receiving emicizumab prophylaxis after Week 24, the timepoints for Arm B (Emi) are expressed relative to first emicizumab dose; baseline for Arm B (Emi) is the same as Week 25 for Arm B (Control).
Time Frame: Baseline and Week 25 (for Arm B (Emi), Study Weeks are relative to first emicizumab dose)
Population: The number analyzed is the number of adolescent participants (12-17 years old) who responded to the questionnaire at baseline and Week 25. Arm D is excluded because no adolescents were enrolled in that arm.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Arm B (Emi): 1.5 mg/kg Emicizumab QW: This arm includes Arm B participants who switched to emicizumab prophylaxis after having completed the first 24 weeks on study with no prophylaxis. After Week 24, emicizumab was administered at a loading dose of 3 mg/kg once a week (QW) subcutaneously (SC) for the first 4 weeks followed by a maintenance dose of 1.5 mg/kg emicizumab QW SC up to the end of study.
Arm/Group | Arm A: 1.5 mg/kg Emicizumab QW | Arm B (Control): No Prophylaxis | Arm B (Emi): 1.5 mg/kg Emicizumab QW | Arm C: 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 4 | 2 | 2 | 26
units on a scale
  Baseline: number analyzed (Participants) | 2 | 2 | 2 | 25
  Baseline | 34.643 (22.728) | 37.143 (12.122) | 30.000 (14.142) | 30.714 (15.625)
  Week 25: number analyzed (Participants) | 3 | 2 | 2 | 22
  Week 25 | 33.095 (17.559) | 30.000 (14.142) | 12.143 (7.071) | 19.286 (14.507)

18. Secondary Outcome: Long-Term Efficacy of Emicizumab: Model-Based Annualized Bleed Rates (ABR) for Treated Bleeds, All Bleeds, Treated Spontaneous Bleeds, Treated Joint Bleeds, and Treated Target Joint Bleeds, All Enrolled Participants
Description: The number of bleeds over the efficacy period was assessed as an ABR using a negative binomial (NB) regression model, which accounts for different follow-up times. Treated bleeds: a bleed for which coagulation factors were administered. All bleeds included both treated and non-treated bleeds. Treated spontaneous bleeds: treated bleeds with no known contributing factor (e.g., trauma, surgery). Treated joint bleeds: treated bleeds in a joint associated with unusual sensation (aura) in a joint, in combination with another symptom: swelling/warmth, pain/decreased range of motion (RoM), or difficulty moving the joint. Treated target joint bleeds: treated joint bleeds in a target joint, defined as a joint in which greater than or equal to (>/=) 3 treated joint bleeds occurred during the last 24 weeks prior to study entry. For all types of bleeds: the 72-hour rule was implemented, and bleeds due to surgery/procedure and bleeds after up-titration were excluded.
Time Frame: From start of emicizumab treatment to study completion (median [min-max] efficacy observation period for all participants: 109.29 [0.1-249.1] weeks)
Population: All enrolled participants; for Arm B, it only includes participants who switched to emicizumab prophylaxis after having completed the first 24 weeks on study with no prophylaxis.
Measure: Number (95% Confidence Interval); unit: bleeds per year
Groups:
- All Participants: 1.5 mg/kg Emicizumab QW: This analysis set included all enrolled participants on the study. For Arm B, it only all participants starting after Week 24 on study when they crossed over to first receive prophylactic treatment with emicizumab. Emicizumab was administered at a loading dose of 3 mg/kg/week SC for the first 4 weeks followed by a maintenance dose of 1.5 mg/kg/week SC up to the end of study. Participants continued to receive bypassing agent therapy to treat breakthrough bleeds, with rFVIIa and/or aPCC.
Arm/Group | Arm A: 1.5 mg/kg Emicizumab QW | Arm B (Emi): 1.5 mg/kg Emicizumab QW | Arm C: 1.5 mg/kg Emicizumab QW | Arm D: 1.5 mg/kg Emicizumab QW | All Participants: 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 35 | 18 | 49 | 11 | 113
bleeds per year
  Treated Bleeds | 1.9 [1.02 to 3.53] | 0.6 [0.22 to 1.36] | 3.2 [1.51 to 6.65] | 1.5 [0.20 to 11.72] | 2.4 [1.50 to 3.82]
  All Bleeds | 3.5 [2.11 to 5.74] | 1.3 [0.66 to 2.39] | 4.3 [2.43 to 7.77] | 2.3 [0.79 to 6.77] | 3.6 [2.55 to 5.13]
  Treated Spontaneous Bleeds | 0.6 [0.33 to 1.26] | 0.1 [0.06 to 0.29] | 2.1 [0.89 to 4.80] | 0.8 [0.07 to 9.16] | 1.3 [0.76 to 2.18]
  Treated Joint Bleeds | 0.5 [0.16 to 1.69] | 0.1 [0.04 to 0.31] | 0.4 [0.14 to 0.96] | 0.4 [0.05 to 3.41] | 0.4 [0.21 to 0.82]
  Treated Target Joint Bleeds | 0.1 [0.01 to 0.31] | 0.01 [0.01 to 0.18] | 0.3 [0.09 to 0.84] | 0.3 [0.04 to 2.36] | 0.2 [0.10 to 0.57]

19. Secondary Outcome: Long-Term Efficacy of Emicizumab: Mean Calculated Annualized Bleed Rates (ABR) for Treated Bleeds, All Bleeds, Treated Spontaneous Bleeds, Treated Joint Bleeds, and Treated Target Joint Bleeds, All Enrolled Participants
Description: as for outcome 10
Time Frame: as for outcome 18
Population: as for outcome 18
Measure: Mean (95% Confidence Interval); unit: bleeds per year
Groups:
- All Participants: 1.5 mg/kg Emicizumab QW: This analysis set included all enrolled participants on the study. For Arm B, it only included participants starting after Week 24 on study when they crossed over to first receive prophylactic treatment with emicizumab. Emicizumab was administered at a loading dose of 3 mg/kg/week SC for the first 4 weeks followed by a maintenance dose of 1.5 mg/kg/week SC up to the end of study. Participants continued to receive bypassing agent therapy to treat breakthrough bleeds, with rFVIIa and/or aPCC.
Arm/Group | Arm A: 1.5 mg/kg Emicizumab QW | Arm B (Emi): 1.5 mg/kg Emicizumab QW | Arm C: 1.5 mg/kg Emicizumab QW | Arm D: 1.5 mg/kg Emicizumab QW | All Participants: 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 35 | 18 | 49 | 11 | 113
bleeds per year
  Treated Bleeds | 2.9 [0.58 to 8.63] | 0.6 [0.00 to 4.85] | 3.3 [0.77 to 9.28] | 1.6 [0.14 to 6.61] | 2.6 [0.46 to 8.16]
  All Bleeds | 4.8 [1.49 to 11.33] | 1.3 [0.07 to 6.11] | 4.6 [1.40 to 11.09] | 2.5 [0.42 to 8.02] | 3.9 [1.05 to 10.13]
  Treated Spontaneous Bleeds | 1.2 [0.06 to 5.99] | 0.2 [0.00 to 4.01] | 2.2 [0.32 to 7.59] | 0.9 [0.01 to 5.33] | 1.5 [0.10 to 6.35]
  Treated Joint Bleeds | 0.9 [0.02 to 5.42] | 0.1 [0.00 to 3.95] | 0.4 [0.00 to 4.53] | 0.4 [0.00 to 4.56] | 0.5 [0.00 to 4.73]
  Treated Target Joint Bleeds | 0.4 [0.00 to 4.44] | 0.1 [0.00 to 3.79] | 0.3 [0.00 to 4.35] | 0.4 [0.00 to 4.40] | 0.3 [0.00 to 4.30]

20. Secondary Outcome: Long-Term Efficacy of Emicizumab: Median Calculated Annualized Bleed Rates (ABR) for Treated Bleeds, All Bleeds, Treated Spontaneous Bleeds, Treated Joint Bleeds, and Treated Target Joint Bleeds, All Enrolled Participants
Description: as for outcome 10
Time Frame: as for outcome 18
Population: as for outcome 18
Measure: Median (Inter-Quartile Range); unit: bleeds per year
Arm/Group | Arm A: 1.5 mg/kg Emicizumab QW | Arm B (Emi): 1.5 mg/kg Emicizumab QW | Arm C: 1.5 mg/kg Emicizumab QW | Arm D: 1.5 mg/kg Emicizumab QW | All Participants: 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 35 | 18 | 49 | 11 | 113
bleeds per year
  Treated Bleeds | 0.3 [0.00 to 2.05] | 0.0 [0.00 to 0.48] | 0.0 [0.00 to 1.13] | 0.0 [0.00 to 0.67] | 0.0 [0.00 to 1.09]
  All Bleeds | 1.9 [0.22 to 5.13] | 0.5 [0.00 to 2.18] | 0.6 [0.00 to 2.25] | 0.5 [0.00 to 4.41] | 0.6 [0.00 to 3.34]
  Treated Spontaneous Bleeds | 0.0 [0.00 to 0.87] | 0.0 [0.00 to 0.24] | 0.0 [0.00 to 0.47] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.51]
  Treated Joint Bleeds | 0.0 [0.00 to 0.24] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00]
  Treated Target Joint Bleeds | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00]

21. Secondary Outcome: Long-Term Efficacy of Emicizumab: Mean Calculated Annualized Bleed Rates (ABR) for Treated Bleeds Per 12-Week Intervals Over Time, All Enrolled Participants
Description: The number of treated bleeds over the efficacy period was calculated as: ABR = (number of bleeds/number of days during the efficacy period) x 365.25. Treated bleeds: a bleed for which coagulation factors were administered. The 72-hour rule was implemented: two bleeds of the same type and at the same anatomical location were counted as one bleed if the second bleed occurred within 72 hours from the last treatment for the first bleed. Bleeds due to surgery/procedure were excluded. For participants whose dose was up-titrated, the efficacy period ended the day before the first day on the up-titrated dose.
Time Frame: 1-12, 13-24, 25-36, 37-48, 49-60, 61-72, 73-84, 85-96, 97-108, 109-120, 121-132, 133-144, 145-156, 157-168, 169-180, 181-192, 193-204, 205-216, 217-228, and 229-240 weeks
Population: All enrolled participants; for Arm B, it only includes participants who switched to emicizumab prophylaxis after having completed the first 24 weeks on study with no prophylaxis. The number analyzed includes participants with available data over each interval.
Measure: Mean (95% Confidence Interval); unit: treated bleeds per year
Arm/Group | All Participants: 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 113
treated bleeds per year
  1 to 12 Weeks: number analyzed (Participants) | 110
  1 to 12 Weeks | 3.9 [1.05 to 10.12]
  13 to 24 Weeks: number analyzed (Participants) | 109
  13 to 24 Weeks | 2.2 [0.31 to 7.53]
  25 to 36 Weeks: number analyzed (Participants) | 102
  25 to 36 Weeks | 0.9 [0.01 to 5.31]
  37 to 48 Weeks: number analyzed (Participants) | 101
  37 to 48 Weeks | 0.3 [0.00 to 4.38]
  49 to 60 Weeks: number analyzed (Participants) | 99
  49 to 60 Weeks | 0.4 [0.00 to 4.56]
  61 to 72 Weeks: number analyzed (Participants) | 98
  61 to 72 Weeks | 0.5 [0.00 to 4.73]
  73 to 84 Weeks: number analyzed (Participants) | 92
  73 to 84 Weeks | 0.6 [0.00 to 4.80]
  85 to 96 Weeks: number analyzed (Participants) | 79
  85 to 96 Weeks | 0.4 [0.00 to 4.46]
  97 to 108 Weeks: number analyzed (Participants) | 67
  97 to 108 Weeks | 0.5 [0.00 to 4.71]
  109 to 120 Weeks: number analyzed (Participants) | 50
  109 to 120 Weeks | 0.0 [NA to 3.69] — The lower limit of the 95% confidence interval could not be calculated because too few events had occurred.
  121 to 132 Weeks: number analyzed (Participants) | 44
  121 to 132 Weeks | 0.4 [0.00 to 4.48]
  133 to 144 Weeks: number analyzed (Participants) | 37
  133 to 144 Weeks | 0.5 [0.00 to 4.62]
  145 to 156 Weeks: number analyzed (Participants) | 31
  145 to 156 Weeks | 0.4 [0.00 to 4.53]
  157 to 168 Weeks: number analyzed (Participants) | 28
  157 to 168 Weeks | 0.2 [0.00 to 4.01]
  169 to 180 Weeks: number analyzed (Participants) | 23
  169 to 180 Weeks | 0.2 [0.00 to 4.08]
  181 to 192 Weeks: number analyzed (Participants) | 19
  181 to 192 Weeks | 0.0 [NA to 3.69] — The lower limit of the 95% confidence interval could not be calculated because too few events had occurred.
  193 to 204 Weeks: number analyzed (Participants) | 13
  193 to 204 Weeks | 0.0 [NA to 3.69] — The lower limit of the 95% confidence interval could not be calculated because too few events had occurred.
  205 to 216 Weeks: number analyzed (Participants) | 9
  205 to 216 Weeks | 0.0 [NA to 3.69] — The lower limit of the 95% confidence interval could not be calculated because too few events had occurred.
  217 to 228 Weeks: number analyzed (Participants) | 4
  217 to 228 Weeks | 0.0 [NA to 3.69] — The lower limit of the 95% confidence interval could not be calculated because too few events had occurred.
  229 to 240 Weeks: number analyzed (Participants) | 2
  229 to 240 Weeks | 0.0 [NA to 3.69] — The lower limit of the 95% confidence interval could not be calculated because too few events had occurred.

22. Secondary Outcome: Long-Term Efficacy of Emicizumab: Median Calculated Annualized Bleed Rates (ABR) for Treated Bleeds Per 12-Week Intervals Over Time, All Enrolled Participants
Description: as for outcome 21
Time Frame: as for outcome 21
Population: as for outcome 21
Measure: Median (Inter-Quartile Range); unit: treated bleeds per year
Arm/Group | All Participants: 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 113
treated bleeds per year
  1 to 12 Weeks: number analyzed (Participants) | 110
  1 to 12 Weeks | 0.0 [0.00 to 4.35]
  13 to 24 Weeks: number analyzed (Participants) | 109
  13 to 24 Weeks | 0.0 [0.00 to 0.00]
  25 to 36 Weeks: number analyzed (Participants) | 102
  25 to 36 Weeks | 0.0 [0.00 to 0.00]
  37 to 48 Weeks: number analyzed (Participants) | 101
  37 to 48 Weeks | 0.0 [0.00 to 0.00]
  49 to 60 Weeks: number analyzed (Participants) | 99
  49 to 60 Weeks | 0.0 [0.00 to 0.00]
  61 to 72 Weeks: number analyzed (Participants) | 98
  61 to 72 Weeks | 0.0 [0.00 to 0.00]
  73 to 84 Weeks: number analyzed (Participants) | 92
  73 to 84 Weeks | 0.0 [0.00 to 0.00]
  85 to 96 Weeks: number analyzed (Participants) | 79
  85 to 96 Weeks | 0.0 [0.00 to 0.00]
  97 to 108 Weeks: number analyzed (Participants) | 67
  97 to 108 Weeks | 0.0 [0.00 to 0.00]
  109 to 120 Weeks: number analyzed (Participants) | 50
  109 to 120 Weeks | 0.0 [0.00 to 0.00]
  121 to 132 Weeks: number analyzed (Participants) | 44
  121 to 132 Weeks | 0.0 [0.00 to 0.00]
  133 to 144 Weeks: number analyzed (Participants) | 37
  133 to 144 Weeks | 0.0 [0.00 to 0.00]
  145 to 156 Weeks: number analyzed (Participants) | 31
  145 to 156 Weeks | 0.0 [0.00 to 0.00]
  157 to 168 Weeks: number analyzed (Participants) | 28
  157 to 168 Weeks | 0.0 [0.00 to 0.00]
  169 to 180 Weeks: number analyzed (Participants) | 23
  169 to 180 Weeks | 0.0 [0.00 to 0.00]
  181 to 192 Weeks: number analyzed (Participants) | 19
  181 to 192 Weeks | 0.0 [0.00 to 0.00]
  193 to 204 Weeks: number analyzed (Participants) | 13
  193 to 204 Weeks | 0.0 [0.00 to 0.00]
  205 to 216 Weeks: number analyzed (Participants) | 9
  205 to 216 Weeks | 0.0 [0.00 to 0.00]
  217 to 228 Weeks: number analyzed (Participants) | 4
  217 to 228 Weeks | 0.0 [0.00 to 0.00]
  229 to 240 Weeks: number analyzed (Participants) | 2
  229 to 240 Weeks | 0.0 [0.00 to 0.00]

23. Secondary Outcome: Long-Term Efficacy of Emicizumab: Mean Calculated Annualized Bleed Rates (ABR) for All Bleeds Per 12-Week Intervals Over Time, All Enrolled Participants
Description: The number of all bleeds over the efficacy period was calculated as: ABR = (number of bleeds/number of days during the efficacy period) x 365.25. All bleeds included both treated bleeds (with coagulation factors) and non-treated bleeds. The 72-hour rule was implemented: two bleeds of the same type and at the same anatomical location were counted as one bleed if the second bleed occurred within 72 hours from the last treatment for the first bleed. Bleeds due to surgery/procedure were excluded. For participants whose dose was up-titrated, the efficacy period ended the day before the first day on the up-titrated dose.
Time Frame: as for outcome 21
Population: as for outcome 21
Measure: Mean (95% Confidence Interval); unit: all bleeds per year
Arm/Group | All Participants: 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 113
all bleeds per year
  1 to 12 Weeks: number analyzed (Participants) | 110
  1 to 12 Weeks | 6.2 [2.35 to 13.40]
  13 to 24 Weeks: number analyzed (Participants) | 109
  13 to 24 Weeks | 3.4 [0.78 to 9.29]
  25 to 36 Weeks: number analyzed (Participants) | 102
  25 to 36 Weeks | 1.5 [0.11 to 6.40]
  37 to 48 Weeks: number analyzed (Participants) | 101
  37 to 48 Weeks | 1.4 [0.09 to 6.29]
  49 to 60 Weeks: number analyzed (Participants) | 99
  49 to 60 Weeks | 1.1 [0.04 to 5.74]
  61 to 72 Weeks: number analyzed (Participants) | 98
  61 to 72 Weeks | 1.0 [0.02 to 5.53]
  73 to 84 Weeks: number analyzed (Participants) | 92
  73 to 84 Weeks | 1.3 [0.07 to 6.12]
  85 to 96 Weeks: number analyzed (Participants) | 79
  85 to 96 Weeks | 1.0 [0.02 to 5.56]
  97 to 108 Weeks: number analyzed (Participants) | 67
  97 to 108 Weeks | 1.2 [0.05 to 5.86]
  109 to 120 Weeks: number analyzed (Participants) | 50
  109 to 120 Weeks | 0.9 [0.01 to 5.34]
  121 to 132 Weeks: number analyzed (Participants) | 44
  121 to 132 Weeks | 0.8 [0.01 to 5.20]
  133 to 144 Weeks: number analyzed (Participants) | 37
  133 to 144 Weeks | 0.5 [0.00 to 4.62]
  145 to 156 Weeks: number analyzed (Participants) | 31
  145 to 156 Weeks | 0.8 [0.01 to 5.29]
  157 to 168 Weeks: number analyzed (Participants) | 28
  157 to 168 Weeks | 0.3 [0.00 to 4.31]
  169 to 180 Weeks: number analyzed (Participants) | 23
  169 to 180 Weeks | 0.8 [0.01 to 5.14]
  181 to 192 Weeks: number analyzed (Participants) | 19
  181 to 192 Weeks | 0.2 [0.00 to 4.15]
  193 to 204 Weeks: number analyzed (Participants) | 13
  193 to 204 Weeks | 0.0 [NA to 3.69] — The lower limit of the 95% confidence interval could not be calculated because too few events had occurred.
  205 to 216 Weeks: number analyzed (Participants) | 9
  205 to 216 Weeks | 0.0 [NA to 3.69] — The lower limit of the 95% confidence interval could not be calculated because too few events had occurred.
  217 to 228 Weeks: number analyzed (Participants) | 4
  217 to 228 Weeks | 0.0 [NA to 3.69] — The lower limit of the 95% confidence interval could not be calculated because too few events had occurred.
  229 to 240 Weeks: number analyzed (Participants) | 2
  229 to 240 Weeks | 0.0 [NA to 3.69] — The lower limit of the 95% confidence interval could not be calculated because too few events had occurred.

24. Secondary Outcome: Long-Term Efficacy of Emicizumab: Median Calculated Annualized Bleed Rates (ABR) for All Bleeds Per 12-Week Intervals Over Time, All Enrolled Participants
Description: as for outcome 23
Time Frame: as for outcome 21
Population: as for outcome 21
Measure: Median (Inter-Quartile Range); unit: all bleeds per year
Arm/Group | All Participants: 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 113
all bleeds per year
  1 to 12 Weeks: number analyzed (Participants) | 110
  1 to 12 Weeks | 0.0 [0.00 to 8.70]
  13 to 24 Weeks: number analyzed (Participants) | 109
  13 to 24 Weeks | 0.0 [0.00 to 4.35]
  25 to 36 Weeks: number analyzed (Participants) | 102
  25 to 36 Weeks | 0.0 [0.00 to 0.00]
  37 to 48 Weeks: number analyzed (Participants) | 101
  37 to 48 Weeks | 0.0 [0.00 to 0.00]
  49 to 60 Weeks: number analyzed (Participants) | 99
  49 to 60 Weeks | 0.0 [0.00 to 0.00]
  61 to 72 Weeks: number analyzed (Participants) | 98
  61 to 72 Weeks | 0.0 [0.00 to 0.00]
  73 to 84 Weeks: number analyzed (Participants) | 92
  73 to 84 Weeks | 0.0 [0.00 to 0.00]
  85 to 96 Weeks: number analyzed (Participants) | 79
  85 to 96 Weeks | 0.0 [0.00 to 0.00]
  97 to 108 Weeks: number analyzed (Participants) | 67
  97 to 108 Weeks | 0.0 [0.00 to 0.00]
  109 to 120 Weeks: number analyzed (Participants) | 50
  109 to 120 Weeks | 0.0 [0.00 to 0.00]
  121 to 132 Weeks: number analyzed (Participants) | 44
  121 to 132 Weeks | 0.0 [0.00 to 0.00]
  133 to 144 Weeks: number analyzed (Participants) | 37
  133 to 144 Weeks | 0.0 [0.00 to 0.00]
  145 to 156 Weeks: number analyzed (Participants) | 31
  145 to 156 Weeks | 0.0 [0.00 to 0.00]
  157 to 168 Weeks: number analyzed (Participants) | 28
  157 to 168 Weeks | 0.0 [0.00 to 0.00]
  169 to 180 Weeks: number analyzed (Participants) | 23
  169 to 180 Weeks | 0.0 [0.00 to 0.00]
  181 to 192 Weeks: number analyzed (Participants) | 19
  181 to 192 Weeks | 0.0 [0.00 to 0.00]
  193 to 204 Weeks: number analyzed (Participants) | 13
  193 to 204 Weeks | 0.0 [0.00 to 0.00]
  205 to 216 Weeks: number analyzed (Participants) | 9
  205 to 216 Weeks | 0.0 [0.00 to 0.00]
  217 to 228 Weeks: number analyzed (Participants) | 4
  217 to 228 Weeks | 0.0 [0.00 to 0.00]
  229 to 240 Weeks: number analyzed (Participants) | 2
  229 to 240 Weeks | 0.0 [0.00 to 0.00]

25. Secondary Outcome: Long-Term Efficacy of Emicizumab: Mean Calculated Annualized Bleed Rates (ABR) for Treated Spontaneous Bleeds Per 12-Week Intervals Over Time, All Enrolled Participants
Description: The number of treated spontaneous bleeds over the efficacy period was calculated as: ABR = (number of bleeds/number of days during the efficacy period) x 365.25. Treated spontaneous bleeds were defined as treated (with coagulation factors) bleeds with no known contributing factor (e.g., trauma, surgery). The 72-hour rule was implemented: two bleeds of the same type and at the same anatomical location were counted as one bleed if the second bleed occurred within 72 hours from the last treatment for the first bleed. Bleeds due to surgery/procedure were excluded. For participants whose dose was up-titrated, the efficacy period ended the day before the first day on the up-titrated dose.
Time Frame: as for outcome 21
Population: as for outcome 21
Measure: Mean (95% Confidence Interval); unit: treated spontaneous bleeds per year
Arm/Group | All Participants: 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 113
treated spontaneous bleeds per year
  1 to 12 Weeks: number analyzed (Participants) | 110
  1 to 12 Weeks | 2.2 [0.31 to 7.56]
  13 to 24 Weeks: number analyzed (Participants) | 109
  13 to 24 Weeks | 1.3 [0.06 to 6.04]
  25 to 36 Weeks: number analyzed (Participants) | 102
  25 to 36 Weeks | 0.4 [0.00 to 4.45]
  37 to 48 Weeks: number analyzed (Participants) | 101
  37 to 48 Weeks | 0.2 [0.00 to 4.04]
  49 to 60 Weeks: number analyzed (Participants) | 99
  49 to 60 Weeks | 0.1 [0.00 to 3.96]
  61 to 72 Weeks: number analyzed (Participants) | 98
  61 to 72 Weeks | 0.2 [0.00 to 4.05]
  73 to 84 Weeks: number analyzed (Participants) | 92
  73 to 84 Weeks | 0.2 [0.00 to 4.08]
  85 to 96 Weeks: number analyzed (Participants) | 79
  85 to 96 Weeks | 0.1 [0.00 to 3.92]
  97 to 108 Weeks: number analyzed (Participants) | 67
  97 to 108 Weeks | 0.3 [0.00 to 4.34]
  109 to 120 Weeks: number analyzed (Participants) | 50
  109 to 120 Weeks | 0.0 [NA to 3.69] — The lower limit of the 95% confidence interval could not be calculated because too few events had occurred.
  121 to 132 Weeks: number analyzed (Participants) | 44
  121 to 132 Weeks | 0.1 [0.00 to 3.89]
  133 to 144 Weeks: number analyzed (Participants) | 37
  133 to 144 Weeks | 0.0 [NA to 3.69] — The lower limit of the 95% confidence interval could not be calculated because too few events had occurred.
  145 to 156 Weeks: number analyzed (Participants) | 31
  145 to 156 Weeks | 0.4 [0.00 to 4.53]
  157 to 168 Weeks: number analyzed (Participants) | 28
  157 to 168 Weeks | 0.2 [0.00 to 4.01]
  169 to 180 Weeks: number analyzed (Participants) | 23
  169 to 180 Weeks | 0.2 [0.00 to 4.08]
  181 to 192 Weeks: number analyzed (Participants) | 19
  181 to 192 Weeks | 0.0 [NA to 3.69] — The lower limit of the 95% confidence interval could not be calculated because too few events had occurred.
  193 to 204 Weeks: number analyzed (Participants) | 13
  193 to 204 Weeks | 0.0 [NA to 3.69] — The lower limit of the 95% confidence interval could not be calculated because too few events had occurred.
  205 to 216 Weeks: number analyzed (Participants) | 9
  205 to 216 Weeks | 0.0 [NA to 3.69] — The lower limit of the 95% confidence interval could not be calculated because too few events had occurred.
  217 to 228 Weeks: number analyzed (Participants) | 4
  217 to 228 Weeks | 0.0 [NA to 3.69] — The lower limit of the 95% confidence interval could not be calculated because too few events had occurred.
  229 to 240 Weeks: number analyzed (Participants) | 2
  229 to 240 Weeks | 0.0 [NA to 3.69] — The lower limit of the 95% confidence interval could not be calculated because too few events had occurred.

26. Secondary Outcome: Long-Term Efficacy of Emicizumab: Median Calculated Annualized Bleed Rates (ABR) for Treated Spontaneous Bleeds Per 12-Week Intervals Over Time, All Enrolled Participants
Description: as for outcome 25
Time Frame: as for outcome 21
Population: as for outcome 21
Measure: Median (Inter-Quartile Range); unit: treated spontaneous bleeds per year
Arm/Group | All Participants: 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 113
treated spontaneous bleeds per year
  1 to 12 Weeks: number analyzed (Participants) | 110
  1 to 12 Weeks | 0.0 [0.00 to 0.00]
  13 to 24 Weeks: number analyzed (Participants) | 109
  13 to 24 Weeks | 0.0 [0.00 to 0.00]
  25 to 36 Weeks: number analyzed (Participants) | 102
  25 to 36 Weeks | 0.0 [0.00 to 0.00]
  37 to 48 Weeks: number analyzed (Participants) | 101
  37 to 48 Weeks | 0.0 [0.00 to 0.00]
  49 to 60 Weeks: number analyzed (Participants) | 99
  49 to 60 Weeks | 0.0 [0.00 to 0.00]
  61 to 72 Weeks: number analyzed (Participants) | 98
  61 to 72 Weeks | 0.0 [0.00 to 0.00]
  73 to 84 Weeks: number analyzed (Participants) | 92
  73 to 84 Weeks | 0.0 [0.00 to 0.00]
  85 to 96 Weeks: number analyzed (Participants) | 79
  85 to 96 Weeks | 0.0 [0.00 to 0.00]
  97 to 108 Weeks: number analyzed (Participants) | 67
  97 to 108 Weeks | 0.0 [0.00 to 0.00]
  109 to 120 Weeks: number analyzed (Participants) | 50
  109 to 120 Weeks | 0.0 [0.00 to 0.00]
  121 to 132 Weeks: number analyzed (Participants) | 44
  121 to 132 Weeks | 0.0 [0.00 to 0.00]
  133 to 144 Weeks: number analyzed (Participants) | 37
  133 to 144 Weeks | 0.0 [0.00 to 0.00]
  145 to 156 Weeks: number analyzed (Participants) | 31
  145 to 156 Weeks | 0.0 [0.00 to 0.00]
  157 to 168 Weeks: number analyzed (Participants) | 28
  157 to 168 Weeks | 0.0 [0.00 to 0.00]
  169 to 180 Weeks: number analyzed (Participants) | 23
  169 to 180 Weeks | 0.0 [0.00 to 0.00]
  181 to 192 Weeks: number analyzed (Participants) | 19
  181 to 192 Weeks | 0.0 [0.00 to 0.00]
  193 to 204 Weeks: number analyzed (Participants) | 13
  193 to 204 Weeks | 0.0 [0.00 to 0.00]
  205 to 216 Weeks: number analyzed (Participants) | 9
  205 to 216 Weeks | 0.0 [0.00 to 0.00]
  217 to 228 Weeks: number analyzed (Participants) | 4
  217 to 228 Weeks | 0.0 [0.00 to 0.00]
  229 to 240 Weeks: number analyzed (Participants) | 2
  229 to 240 Weeks | 0.0 [0.00 to 0.00]

27. Secondary Outcome: Safety Summary of the Overall Number and Percentage of Participants With at Least One Adverse Event, Severity Assessed According to the WHO Toxicity Grading Scale
Description: Investigators sought information on adverse events (AEs) at each contact with participants. The WHO toxicity grading scale was used for assessing AE severity (i.e., intensity of an AE); any AEs not specifically listed in the WHO toxicity grading scale were assessed for severity according to the following grades: Grade 1 is mild; Grade 2 is moderate, Grade 3 is severe; Grade 4 is life-threatening; and Grade 5 is death. Regardless of severity, some AEs may have also met seriousness criteria. The terms "severe" and "serious" are not synonymous; severity and seriousness were independently assessed for each AE. For participants whose emicizumab dose was up-titrated, only data before up-titration is included. aPCC = activated prothrombin complex concentrate; Hypersens.= hypersensitivity
Time Frame: From Baseline until study completion (median [min-max] safety observation period for all participants: 133.97 [0.1-249.1] weeks)
Population: Safety Population: All treated participants grouped by their assigned treatment. For Arm B, data collected while receiving episodic bypassing agents (no prophyalxis) for the first 24 weeks and 1.5 mg/kg emicizumab QW after Week 24 are reported separately under 'Arm B (Control): No Prophylaxis' and 'Arm B (Emi): 1.5 mg/kg Emicizumab QW', respectively.
Measure: Count of Participants; unit: Participants
Groups:
- Arm B (Emi): 1.5 mg/kg Emicizumab QW: This arm includes Arm B participants who switched to emicizumab prophylaxis after completing at least 24-week no prophylaxis. Emicizumab was administered at a loading dose of 3 mg/kg/week SC for the first 4 weeks (after at least 24 weeks) followed by a maintenance dose of 1.5 mg/kg/week SC up to the end of study. Data reported represents data collected during emicizumab treatment only.
Arm/Group | Arm A: 1.5 mg/kg Emicizumab QW | Arm B (Control): No Prophylaxis | Arm B (Emi): 1.5 mg/kg Emicizumab QW | Arm C: 1.5 mg/kg Emicizumab QW | Arm D: 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 34 | 18 | 18 | 49 | 11
Participants
  Any Adverse Event (AE) | 34 | 9 | 15 | 46 | 9
  AE with Fatal Outcome | 0 | 0 | 0 | 1 | 0
  Serious AE | 10 | 4 | 4 | 9 | 2
  AE Leading to Withdrawal from Treatment | 2 | 0 | 0 | 1 | 0
  AE Leading to Dose Mod./Interruption | 1 | 0 | 0 | 5 | 0
  Grade ≥3 AE | 10 | 4 | 3 | 7 | 3
  Related AE | 15 | 0 | 4 | 13 | 4
  Local Injection Site Reaction | 9 | 0 | 3 | 7 | 4
  Systemic Hypersens./Anaphylac(tic/toid) Reaction | 0 | 0 | 0 | 0 | 0
  Thrombotic Microangiopathy (TMA) | 1 | 0 | 0 | 2 | 0
  TMA Event Related to aPCC and Emicizumab | 1 | 0 | 0 | 2 | 0
  Thromboembolic Event (TE) | 1 | 1 | 1 | 1 | 0
  TE Event Related to aPCC and Emicizumab | 1 | 0 | 0 | 1 | 0

28. Secondary Outcome: Number of Participants Testing Negative or Positive for the Presence of Anti-Drug Antibodies (ADAs), Including Neutralizing ADAs, During the Study
Description: 'Total ADA Negative' is the sum of all subjects who tested negative for ADA in the 2 following categories: 'ADA Negative', those who are pre-dose ADA negative or are missing pre-dose ADA data and who have all negative post-dose ADA results; and 'ADA Negative (Treatment Unaffected)', a subset who are pre-dose ADA positive but do not have a ≥4-fold increase in post-dose ADA levels compared to baseline measurement. 'Total ADA Positive' is the sum of all subjects who tested positive for ADA in the 2 following categories: 'ADA Positive (Treatment Boosted)', those who are pre-dose ADA positive and have a ≥4-fold increase in post-dose ADA levels compared to baseline measurement; and 'ADA Positive (Treatment Induced)', those who are pre-dose ADA negative or missing data and who have at least one post-dose ADA positive sample. ADA-positive samples were further analyzed for neutralizing capacity using a modified FVIII chromogenic assay; if also positive, they were considered neutralizing ADAs.
Time Frame: as for outcome 27
Population: All emicizumab-treated participants included Arms A, C, and D and Arm B participants who switched to receive emicizumab (Arm B Emi). The overall number of participants analyzed is the number of participants with at least one post-baseline anti-drug antibody assessment.
Measure: Count of Participants; unit: Participants
Groups:
- Arm B (Emi): 1.5 mg/kg Emicizumab QW: This arm includes Arm B participants who switched to emicizumab prophylaxis after completing at least 24-week no prophylaxis. Emicizumab was administered at a loading dose of 3 mg/kg/week SC for the first 4 weeks (after at least 24 weeks) followed by a maintenance dose of 1.5 mg/kg/week SC up to the end of study.
Arm/Group | Arm A: 1.5 mg/kg Emicizumab QW | Arm B (Emi): 1.5 mg/kg Emicizumab QW | Arm C: 1.5 mg/kg Emicizumab QW | Arm D: 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 33 | 18 | 49 | 11
Participants
  Total ADA Negative (Neg+Neg Unaffected) | 33 | 18 | 47 | 11
  ADA Negative, Negative | 33 | 17 | 46 | 11
  ADA Negative, Negative (Treatment Unaffected) | 0 | 1 | 1 | 0
  Total ADA Positive (Boosted + Induced) | 0 | 0 | 2 | 0
  ADA Positive, Positive (Treatment Boosted) | 0 | 0 | 0 | 0
  ADA Positive, Positive (Treatment Induced) | 0 | 0 | 2 | 0
  ADA Positive with Neutralizing ADAs | 0 | 0 | 2 | 0

29. Secondary Outcome: Plasma Trough Concentrations of Emicizumab at Specified Timepoints
Description: Plasma concentrations of emicizumab were analyzed using a validated Enzyme Linked Immunosorbent Assay (ELISA). The lower limit of quantification (LLOQ) was 100 nanograms per milliliter (ng/mL). Because participants in Arm B switched from episodic bypassing agents to start receiving emicizumab prophylaxis after Week 24, the timepoints for Arm B (Emi) are expressed relative to first emicizumab dose.
Time Frame: Pre-dose (0 hour [hr]) on Weeks 1-5, 7, 9, 13, 17, 21, 25, 33, 41, 49, 61, 73, 85, 97, 109, 121, 133, 145, 157, and 169 (For Arm B (Emi), Study Weeks are relative to first emicizumab dose)
Population: Pharmacokinetic (PK) evaluable population included all participants who received at least one dose of emicizumab and had at least one post-dose emicizumab concentration result. The number analyzed includes participants with PK samples at each timepoint.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (mcg/mL)
Arm/Group | Arm A: 1.5 mg/kg Emicizumab QW | Arm B (Emi): 1.5 mg/kg Emicizumab QW | Arm C: 1.5 mg/kg Emicizumab QW | Arm D: 1.5 mg/kg Emicizumab QW | All Participants: 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 34 | 18 | 49 | 11 | 112
micrograms per milliliter (mcg/mL)
  Week 1: number analyzed (Participants) | 33 | 18 | 48 | 11 | 110
  Week 1 | NA (NA) — No data available because all of the measurements were below the LLOQ. | NA (NA) — No data available because all of the measurements were below the LLOQ. | NA (NA) — No data available because all of the measurements were below the LLOQ. | NA (NA) — No data available because all of the measurements were below the LLOQ. | NA (NA) — No data available because all of the measurements were below the LLOQ.
  Week 2: number analyzed (Participants) | 34 | 17 | 46 | 10 | 107
  Week 2 | 16.2 (4.4) | 21.7 (10.6) | 15.8 (5.5) | 18.3 (6.5) | 17.1 (6.6)
  Week 3: number analyzed (Participants) | 34 | 18 | 47 | 11 | 110
  Week 3 | 31.6 (7.3) | 32.3 (10.4) | 31.7 (8.3) | 32.7 (13.0) | 31.9 (8.8)
  Week 4: number analyzed (Participants) | 32 | 18 | 46 | 11 | 107
  Week 4 | 43.8 (12.2) | 44.6 (18.6) | 44.7 (11.5) | 49.0 (13.5) | 44.9 (13.2)
  Week 5: number analyzed (Participants) | 33 | 18 | 46 | 11 | 108
  Week 5 | 53.5 (15.1) | 52.2 (14.2) | 54.0 (13.2) | 59.1 (14.6) | 54.1 (14.0)
  Week 7: number analyzed (Participants) | 33 | 17 | 46 | 11 | 107
  Week 7 | 52.8 (16.2) | 53.3 (18.0) | 53.6 (14.3) | 54.9 (9.2) | 53.4 (14.9)
  Week 9: number analyzed (Participants) | 32 | 17 | 46 | 11 | 106
  Week 9 | 50.4 (12.4) | 48.9 (16.7) | 52.6 (15.7) | 53.7 (13.8) | 51.5 (14.7)
  Week 13: number analyzed (Participants) | 32 | 17 | 46 | 11 | 106
  Week 13 | 49.3 (13.4) | 45.2 (16.2) | 52.6 (15.0) | 53.4 (14.0) | 50.5 (14.7)
  Week 17: number analyzed (Participants) | 32 | 17 | 46 | 11 | 106
  Week 17 | 50.7 (15.0) | 46.5 (17.4) | 51.2 (14.9) | 57.5 (16.9) | 51.0 (15.6)
  Week 21: number analyzed (Participants) | 32 | 17 | 44 | 11 | 104
  Week 21 | 52.6 (17.4) | 44.5 (15.4) | 51.6 (17.1) | 55.0 (13.7) | 51.1 (16.6)
  Week 25: number analyzed (Participants) | 31 | 17 | 45 | 11 | 104
  Week 25 | 54.6 (19.1) | 45.8 (18.6) | 50.4 (16.8) | 52.8 (14.1) | 51.2 (17.6)
  Week 33: number analyzed (Participants) | 27 | 17 | 41 | 10 | 95
  Week 33 | 50.7 (17.2) | 48.1 (21.1) | 54.8 (16.7) | 57.1 (15.2) | 52.7 (17.5)
  Week 41: number analyzed (Participants) | 27 | 17 | 40 | 10 | 94
  Week 41 | 45.3 (13.7) | 49.3 (25.9) | 54.8 (23.4) | 63.3 (19.4) | 52.0 (21.6)
  Week 49: number analyzed (Participants) | 27 | 15 | 40 | 9 | 91
  Week 49 | 48.0 (12.3) | 54.6 (27.6) | 56.1 (22.2) | 55.1 (18.7) | 53.3 (20.5)
  Week 61: number analyzed (Participants) | 27 | 15 | 40 | 10 | 92
  Week 61 | 52.2 (16.3) | 51.8 (33.4) | 60.9 (27.7) | 53.2 (13.8) | 56.0 (24.8)
  Week 73: number analyzed (Participants) | 27 | 12 | 39 | 9 | 87
  Week 73 | 55.5 (14.9) | 45.6 (26.2) | 62.9 (24.9) | 51.9 (13.0) | 57.1 (22.0)
  Week 85: number analyzed (Participants) | 27 | 10 | 36 | 5 | 78
  Week 85 | 56.9 (18.3) | 42.5 (34.4) | 56.6 (22.7) | 50.9 (12.5) | 54.5 (22.7)
  Week 97: number analyzed (Participants) | 25 | 9 | 27 | 5 | 66
  Week 97 | 53.2 (15.2) | 34.4 (26.4) | 54.6 (20.0) | 53.8 (16.9) | 51.3 (19.9)
  Week 109: number analyzed (Participants) | 23 | 6 | 15 | 3 | 47
  Week 109 | 49.6 (15.9) | 32.8 (31.4) | 47.4 (12.4) | 49.3 (12.8) | 46.7 (17.6)
  Week 121: number analyzed (Participants) | 19 | 7 | 11 | 2 | 39
  Week 121 | 53.8 (16.3) | 36.1 (33.6) | 46.3 (12.5) | 53.1 (5.0) | 48.5 (19.7)
  Week 133: number analyzed (Participants) | 15 | 6 | 7 | 1 | 29
  Week 133 | 50.5 (15.9) | 48.7 (29.4) | 49.0 (18.5) | 52.0 (NA) — Standard deviation (SD) could not be calculated for single participant data. | 49.8 (18.8)
  Week 145: number analyzed (Participants) | 13 | 4 | 5 | 2 | 24
  Week 145 | 51.3 (16.6) | 38.2 (19.0) | 44.0 (21.7) | 49.5 (10.3) | 47.4 (17.4)
  Week 157: number analyzed (Participants) | 15 | 0 | 4 | 2 | 21
  Week 157 | 58.0 (16.5) |  | 45.5 (17.0) | 55.4 (19.2) | 55.3 (16.7)
  Week 169: number analyzed (Participants) | 12 | 0 | 3 | 1 | 16
  Week 169 | 55.0 (19.3) |  | 43.2 (20.2) | 50.8 (NA) — Standard deviation (SD) could not be calculated for single participant data. | 52.5 (18.7)

ADVERSE EVENTS:
Time Frame: From Baseline until study completion (median [min-max] safety observation period for all participants: 133.97 [0.1-249.1] weeks)
Description: Safety Population: All treated subjects grouped by treatment (including after up-titration). For Arm B, data collected with episodic bypassing agents (no prophyalxis) for first 24 weeks and with 1.5 mg/kg emicizumab QW after Week 24 are reported separately under Arm B (Control): No Prophylaxis and Arm B (Emi): 1.5 mg/kg Emicizumab QW, respectively.
Groups:
- Arm B (Control): No Prophylaxis: Participants who were receiving episodic treatment with bypassing agents prior to study entry and were randomized to study Arm B continued with their prior episodic treatment regimen for the first 24 weeks of the study; they did not receive emicizumab prophylaxis during that time. The safety data reported here represents data collected from all Arm B participants during the first 24 weeks of 'no prophylaxis'; safety data from Arm B participants who switched to emicizumab after Week 24 are reported separately under Arm B (Emi): 1.5 mg/kg Emicizumab QW.
Arm/Group | Arm A: 1.5 mg/kg Emicizumab QW | Arm B (Control): No Prophylaxis | Arm B (Emi): 1.5 mg/kg Emicizumab QW | Arm C: 1.5 mg/kg Emicizumab QW | Arm D: 1.5 mg/kg Emicizumab QW
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/18 | 0/18 | 1/49 | 0/11
Serious Adverse Events (participants affected / at risk) | 11/34 | 5/18 | 4/18 | 9/49 | 2/11
Other Adverse Events (participants affected / at risk) | 33/34 | 9/18 | 15/18 | 42/49 | 9/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: 1.5 mg/kg Emicizumab QW (N=34) | Arm B (Control): No Prophylaxis (N=18) | Arm B (Emi): 1.5 mg/kg Emicizumab QW (N=18) | Arm C: 1.5 mg/kg Emicizumab QW (N=49) | Arm D: 1.5 mg/kg Emicizumab QW (N=11)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombophlebitis superficial (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 1 (1) | 2 (3) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cavernous sinus thrombosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Soft tissue haemorrhage (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth development disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Meningitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vascular device infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device related sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Device loosening (Product Issues) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intentional self-injury (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subcapsular renal haematoma (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: 1.5 mg/kg Emicizumab QW (N=34) | Arm B (Control): No Prophylaxis (N=18) | Arm B (Emi): 1.5 mg/kg Emicizumab QW (N=18) | Arm C: 1.5 mg/kg Emicizumab QW (N=49) | Arm D: 1.5 mg/kg Emicizumab QW (N=11)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Enteritis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 4 (4) | 0 (0) | 2 (2) | 2 (3) | 2 (2)
Chest pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 3 (4) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Injection site reaction (General disorders) | 9 (18) | 0 (0) | 3 (3) | 8 (21) | 4 (5)
Pyrexia (General disorders) | 2 (2) | 1 (1) | 2 (2) | 8 (10) | 1 (1)
Folliculitis (Infections and infestations) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 11 (29) | 2 (2) | 7 (14) | 16 (27) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 8 (21) | 2 (2) | 2 (2) | 7 (8) | 2 (2)
Post procedural constipation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural hypotension (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural nausea (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (17) | 0 (0) | 6 (9) | 12 (33) | 3 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 6 (9) | 1 (1) | 4 (4) | 13 (22) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Dental caries (Gastrointestinal disorders) | 2 (3) | 0 (0) | 3 (4) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 0 (0) | 1 (1) | 5 (8) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (5) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device related thrombosis (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Influenza (Infections and infestations) | 1 (2) | 0 (0) | 2 (2) | 10 (10) | 0 (0)
Gastroenteritis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Incision site swelling (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Skin laceration (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 3 (4) | 1 (1)
Body temperature increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Indeterminable ABO blood type (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Prothrombin fragment 1.2 increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device occlusion (Product Issues) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 5 (5) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hand dermatitis (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neurodermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.